CLINICAL TRIAL: NCT03135405
Title: Controlling Hypertension in Native American and Other Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: American Heart Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Emily Schroeder, Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CO-16-2400; 2P30DK092923 (NIH); K23DK099237 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Automated messages; Behavioral: Home BP monitors; Behavioral: Care partner reminders

INTERVENTIONS:
Behavioral: Automated messages — Automated motivational messages and visit and medication reminders will be provided via interactive voice response calls or text messages.
  Arms: Intervention
Behavioral: Home BP monitors — Participants will have the option of receiving home blood pressure monitors.
  Arms: Intervention
Behavioral: Care partner reminders — Participants will have the option of designating a care partner who will also receive automated reminder calls or text messages.
  Arms: Intervention

SUMMARY:
The study evaluates the use of automated motivational messages, visit reminders, and medication reminders (using interactive voice response technology or text messages) to improve blood pressure control among adults with hypertension that receive their care at the First Nations Community Healthsource clinic in Albuquerque, New Mexico. Half of the participants will receive usual care, while the other half will receive the automated calls or text messages and have the option to receive home blood pressure monitors and/or designate a care partner who will also receive messages. Participants will be followed for 12 months.

DETAILED DESCRIPTION:
American Indians and Alaskan Natives (AI/ANs) face pervasive health disparities in comparison to other racial and ethnic groups in the United States. Treatment of hypertension is a pillar of cardiovascular disease prevention. Hypertension is the most common chronic health condition in the U.S. Uncontrolled hypertension increases the risk of acute myocardial infarction, stroke, kidney failure, and congestive heart failure. Hypertension rates are high, levels of control are low, and disparities in care are evident in AI/AN populations.

This study will take place at First Nations Community Healthsource (FNCH) in Albuquerque, New Mexico. FNCH provides primary medical care to urban AI/AN and other socially disadvantaged residents of the Albuquerque, New Mexico area. Approximately 40% of FNCH clients are AI/AN; Diné (Navajo) is the most common tribal affiliation. Many other clients served by FNCH are undocumented immigrants. Housing insecurity and homelessness are common.

This study will use a FNCH hypertension registry to identify all clients with hypertension (regardless of race or ethnicity). From this group, the study will recruit 512 clients, and randomize the participants without stratification to receive automated messages using an interactive voice recognition and text message intervention or to continue in usual care. Consistent with the principles of pragmatic randomized clinical trials, the study has few exclusion criteria in order to maximize inclusion of clients and generalizability of findings. Potentially eligible clients will be contacted by letter and phone. Those who express interest will complete a baseline visit where they provide informed consent, complete a baseline survey, and have blood pressure measured. The participants will then be randomized either to the intervention or usual care arms. Individuals randomized to the intervention arm will receive: reminders of upcoming appointments at FNCH; requests to reschedule missed appointments; reminders to refill medications; and weekly motivational messages to encourage self-care, appointment keeping, and medication-taking for hypertension. These participants will be offered a home blood pressure monitor and trained to use it if they accept, and will be asked if they wish to nominate a care partner to also receive notices of upcoming and missed appointments. In additional to their usual visits at FNCH, all participants will complete research visits with our study coordinators at 6 and 12 months, where they will again have BP measured and complete brief surveys.

ELIGIBILITY:
Inclusion Criteria:

* At least two prior visits to First Nations Community Healthsource with blood pressure measurements, with at least one visit in the 24 months prior
* Hypertension
* Between ages 21-79

Exclusion Criteria:

* Another preferred site of primary care
* Significant impairment of vision and hearing
* Life-limiting illness
* Renal dialysis
* Receipt of home health care, hospice services or residence in a nursing home
* Dementia
* Pregnancy
* Current incarceration
* Homeless
* No land line or cellular phone access

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 12-months
  Change in systolic blood pressure from baseline

SECONDARY OUTCOMES:
Diastolic blood pressure | 12-months
  Change in diastolic blood pressure from baseline
Medication adherence | 12-months
  Self-reported medication adherence using the Voils instrument
Visit adherence | 12-months
  Proportion of scheduled appointments that are kept, missed or cancelled

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Schroeder, MD, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- First National Community Healthsource, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroeder EB, Moore KR, Manson SM, Baldwin MA, Goodrich GK, Malone AS, Pieper LE, Xu S, Fort MP, Son-Stone L, Johnson D, Steiner JF. A randomized clinical trial of an interactive voice response and text message intervention for individuals with hypertension. J Clin Hypertens (Greenwich). 2020 Jul;22(7):1228-1238. doi: 10.1111/jch.13909. Epub 2020 Jun 9. PMID 32516486
- [Derived] Schroeder EB, Moore K, Manson SM, Baldwin MA, Goodrich GK, Malone AS, Pieper LE, Xu S, Fort MM, Johnson D, Son-Stone L, Steiner JF. An Interactive Voice Response and Text Message Intervention to Improve Blood Pressure Control Among Individuals With Hypertension Receiving Care at an Urban Indian Health Organization: Protocol and Baseline Characteristics of a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2019 Apr 2;8(4):e11794. doi: 10.2196/11794. PMID 30938688